CLINICAL TRIAL: NCT00881764
Title: Anesthesia Exposure and Neurodevelopment in Infants and Children: Pediatric Anesthesia & NeuroDevelopment (PANDA) Study
Brief Title: PANDA (Pediatric Anesthesia & NeuroDevelopment Assessment) Study
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Office of Acquisitions and Grants Services (OAGS) (Unknown)
Responsible Party: Principal Investigator, Lena S. Sun, Emanuel M. Papper Professor of Anesthesiology and Professor of Pediatrics, Columbia University
Other Study IDs: AAAC8756; R34HD060741 (NIH); HHSF223200810036C (Other Grant/Funding Number: DHHS/FDA/OAGS/DCGM); SmartTots (Other: SmartTots)
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Cognition - Other
Keywords: Anesthesia; New York; Columbia; Children; Neurodevelopment; Child development; Pediatric
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed Cohort: Children who had inguinal hernia surgery and general anesthesia before 36 months of age (n=500). These children should be ages 8 yr, 0 mo to 15 yr, 0 mo at the time of the study period.
  Interventions: Procedure: Inguinal hernia surgery; Procedure: General anesthesia
- Unexposed Cohort: Children who are siblings of the exposed children (inguinal hernia surgery and general anesthesia) and differ in age from the exposed children by less than 36 months and have no history of surgery or exposure to volatile and intravenous anesthetics or sedatives including barbiturates, benzodiazepines and chloral hydrate less than 36 months of age. These children should also be ages 8 yr, 0 mo to 15 yr, 0 mo at the time of the study period.

INTERVENTIONS:
Procedure: Inguinal hernia surgery — Non-experimental procedure
  Groups: Exposed Cohort
Procedure: General anesthesia — Non-experimental procedure/treatment
  Groups: Exposed Cohort

SUMMARY:
The purpose of this study is to determine whether the use of anesthetic agents in infants and children have long term adverse effects on neurocognitive development. According to the National Hospital Discharge Survey, around 2.5 million children have surgical procedures requiring anesthesia each year in the US. Recent animal studies have suggested that the exposure of the immature organism to a variety of commonly used anesthetic agents may lead to neurobehavioral functional deficits in vivo and to neuronal apoptosis in vitro. While the relevance of these findings on children exposed to anesthetics remains to be determined, it is clearly critically important to public health that this issue is resolved quickly and clearly.

Hypothesis: Exposure to anesthetic agents within the first three years of life will not significantly impair cognitive functions at ages 8 yr, 0 mo to 15 yr, 0 mo.

DETAILED DESCRIPTION:
The purpose of our study is to compare neurocognitive functions in sibling pairs: one of whom had exposure to anesthesia during surgery before 36 months of age (exposed sibling cohorts) and who would be from ages 8yr, 0 mo to15 yr, 0 mo at the time of the study; and the other who never had anesthesia or surgery less than 36 months of age, is from ages 8yr, 0mo to 15 yr, 0 mo at the time of the study, and is within 36 months of age range from the exposed sibling(unexposed sibling cohort).

Neuropsychological assessments are administered to the sibling cohorts prospectively and parents of the siblings will complete parental interviews/questionnaires. We assess individually neurocognitive, behavioral and emotional function for both exposed and unexposed siblings. Family function will also be evaluated. We will also obtain complete medical history for each participant, including significant perinatal events and social history. We also review medical records when appropriate.

All testing are performed during a one day site visit.

ELIGIBILITY:
Inclusion Criteria:

Exposed cohort:

1. Subjects who had inguinal hernia surgery before 36 months of age
2. Ages 8 yr, 0 mo to 15 yr, 0 mo
3. Gestation age greater or equal to 36 weeks
4. Categorized as ASA I or ASA II
5. English speaking
6. Biologically related to the unexposed sibling

Unexposed cohort:

1. Sibling within 36 months of age of the exposed cohort
2. Never had surgery or exposure to anesthesia prior to 36 months of age
3. Ages 8 yr, 0 mo to 15 yr, 0 mo
4. Gestation age greater or equal to 36 weeks
5. Categorized as ASA I or ASA II

5. English speaking 6. Biologically related to the exposed sibling

Exclusion criteria:

Exposed cohort:

1. Gestational age less than 36 weeks at birth
2. No exposure to surgery or anesthesia prior to 36 months of age
3. Surgery/Anesthesia other than index hernia repair prior to 36 months of age
4. Not categorized as ASA I or ASA II
5. Not ages 8 yr, 0 mo to 15 yr, 0 mo
6. Not English speaking
7. Not biologically related to the unexposed sibling

Unexposed cohort:

1. Gestational age under 36 weeks at birth
2. Any exposure to surgery or anesthesia prior to 36 months of age
3. Not categorized as ASA I or ASA II
4. Not ages 8 yr, 0 mo to 15 yr, 0 mo
5. Not English speaking
6. Not biologically related to the unexposed sibling

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be a multi-center study based at Columbia University with the following participating centers: Boston Children's (Harvard University), Children's Hospital of Philadelphia (University of Pennsylvania), Monroe Carell Children's Hospital (Vanderbilt University), and Morgan Stanley Children's Hospital of New York (Columbia University). Children exposed to anesthesia prior to 36 months must be ages 8 yr, 0 mo to 15 yr, 0 mo and have a sibling with no history of surgery or anesthesia prior to 36 months of age.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2009-05; Primary Completion 2015-04 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in neurocognitive function | Varies; when the participant is 8-15 years of age
  Global cognitive function: verbal, performance and full IQ assessed by Wechsler Abbreviated Scale of Intelligence (WASI). These are one unit of measure for IQ.

SECONDARY OUTCOMES:
Change in domain-specific function related to visual memory and learning | Varies; when the participant is 8-15 years of age
  NEPSY II (A Developmental Neuropsychological Assessment) assesses visual memory learning
Change in domain-specific function related to verbal memory and learning | Varies; when the participant is 8-15 years of age
  California Verbal Learning Test-Children (CVLT-C) assesses verbal memory and learning.
Change in domain-specific function related to receptive language | Varies; when the participant is 8-15 years of age
  NEPSY II (A Developmental Neuropsychological Assessment) is used to assess receptive language and speeded naming.
Change in domain-specific function related to expressive language | Varies; when the participant is 8-15 years of age
  WASI is used to assess expressive language and verbal reasoning
Change in domain-specific function related to working memory | Varies; when the participant is 8-15 years of age
  Weschler Intelligence Scale for Children (WISC-IV) is used to assess working memory, attention and executive function.
Change in domain-specific function related to all executive function components | Varies; when the participant is 8-15 years of age
  Behavior Rating In Executive Function (BRIEF) is used to assess all components of executive function.
Change in domain-specific function related to selective attention and impulsivity | Varies; when the participant is 8-15 years of age
  Continuous Performance Test-II (CPT-II) is used to assess sustained and selective attention as well as impulsivity.
Change in domain-specific function related to cognitive flexibility aspects of executive function | Varies; when the participant is 8-15 years of age
  Delis-Kaplan Executive Function System (DKEFS) is used to assess cognitive flexibility.
Change in domain-specific function related to motor and processing speed | Varies; when the participant is 8-15 years of age
  Grooved pegboard and Weschler Intelligence Scale for Children (WISC-IV) are used to assess motor and processing speed
Changes in behavior | Varies; when the participant is 8-15 years of age
  Childhood Behavior Check List (CBCL) assesses emotionally reactive, anxious/depressed, somatic complaints, withdrawn, attention problems and aggressive behavior.
Changes in adaptive behavior | Varies; when the participant is 8-15 years of age
  Adaptive behavior is assessed using Adaptive Behavior Assessment Systems II (ABAS-II), which measures overall adaptive behavior and skills.
Changes in parental relationships | Varies; when the participant is 8-15 years of age
  Parent Relationship Questionnaire (PRQ) is used to explore parents' perspectives on parent-child relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Lena S Sun, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Children's Hospital Boston, Boston, Massachusetts
  - Columbia University, 622 W. 168th St., New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ikonomidou C, Bosch F, Miksa M, Bittigau P, Vockler J, Dikranian K, Tenkova TI, Stefovska V, Turski L, Olney JW. Blockade of NMDA receptors and apoptotic neurodegeneration in the developing brain. Science. 1999 Jan 1;283(5398):70-4. doi: 10.1126/science.283.5398.70. PMID 9872743
- [Background] Anand KJ, Soriano SG. Anesthetic agents and the immature brain: are these toxic or therapeutic? Anesthesiology. 2004 Aug;101(2):527-30. doi: 10.1097/00000542-200408000-00033. No abstract available. PMID 15277935
- [Background] Anand KJ. Anesthetic neurotoxicity in newborns: should we change clinical practice? Anesthesiology. 2007 Jul;107(1):2-4. doi: 10.1097/01.anes.0000268484.05444.35. No abstract available. PMID 17585205
- [Background] Olney JW, Young C, Wozniak DF, Jevtovic-Todorovic V, Ikonomidou C. Do pediatric drugs cause developing neurons to commit suicide? Trends Pharmacol Sci. 2004 Mar;25(3):135-9. doi: 10.1016/j.tips.2004.01.002. No abstract available. PMID 15019268
- [Background] Walden M, Carrier CT. Sleeping beauties: the impact of sedation on neonatal development. J Obstet Gynecol Neonatal Nurs. 2003 May-Jun;32(3):393-401. doi: 10.1177/0884217503253454. PMID 12774882
- [Background] Mellon RD, Simone AF, Rappaport BA. Use of anesthetic agents in neonates and young children. Anesth Analg. 2007 Mar;104(3):509-20. doi: 10.1213/01.ane.0000255729.96438.b0. PMID 17312200
- [Background] Jevtovic-Todorovic V, Hartman RE, Izumi Y, Benshoff ND, Dikranian K, Zorumski CF, Olney JW, Wozniak DF. Early exposure to common anesthetic agents causes widespread neurodegeneration in the developing rat brain and persistent learning deficits. J Neurosci. 2003 Feb 1;23(3):876-82. doi: 10.1523/JNEUROSCI.23-03-00876.2003. PMID 12574416
- [Background] Slikker et al. FDA science 2005 Forum
- [Background] Slikker W Jr, Zou X, Hotchkiss CE, Divine RL, Sadovova N, Twaddle NC, Doerge DR, Scallet AC, Patterson TA, Hanig JP, Paule MG, Wang C. Ketamine-induced neuronal cell death in the perinatal rhesus monkey. Toxicol Sci. 2007 Jul;98(1):145-58. doi: 10.1093/toxsci/kfm084. Epub 2007 Apr 10. PMID 17426105
- [Background] Olney at al. FDA symposium. 2002:12:488-498
- [Background] Jevtovic-Todorovic V. General anesthetics and the developing brain: friends or foes? J Neurosurg Anesthesiol. 2005 Oct;17(4):204-6. doi: 10.1097/01.ana.0000178111.26972.16. No abstract available. PMID 16184065